CLINICAL TRIAL: NCT06278870
Title: Disitamab Vedotin in Combination With Pyrotinib Versus THP in the First-line Treatment for HER2-positive Advanced Breast Cancer, a Multicentre, Randomized, Double-blind Controlled, Phase III Trial
Brief Title: Disitamab Vedotin + Pyrotinib Versus THP in the First-line Treatment for HER2+ Advanced Breast Cancer Clinical Trial
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYSKY-2023-431-02
Record Dates: First submitted 2023-08-07; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: HER2-positive Metastatic Breast Cancer; First-line Treatment
MeSH Terms: interventions — disitamab vedotin; RC48 antibody; pyrotinib; Trastuzumab; pertuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- disitamab vedotin in combination with pyrotinib (Experimental): disitamab vedotin 2mg/kg IV every 14 days + Pyrotinib 400mg PO daily, with each 28-day cycle. After 6-8 cycles, adding Trastuzumab initially at 8mg/kg IV followed by 6mg/kg IV every 21 days + Pyrotinib 400mg PO daily for maintenance.
  Interventions: Drug: disitamab vedotin; Drug: Pyrotinib; Drug: trastuzumab
- taxane drug in combination with trastuzumab and pertuzumab (Active Comparator): taxane drug (Docetaxel/Paclitaxel/Albumin Paclitaxel/Liposomal Paclitaxel, dosing and administration per latest National Comprehensive Cancer Network(NCCN) and Chinese Society of Clinical Oncology(CSCO) breast cancer guidelines) + Trastuzumab initially at 8mg/kg IV followed by 6mg/kg IV every 21 days + Pertuzumab initially at 840mg IV followed by 420mg IV every 21 days, with each 21-day cycle. After 6-8 cycles, continuing with Trastuzumab at 6mg/kg IV every 21 days + Pertuzumab at 420mg IV every 21 days for maintenance.
  Interventions: Drug: trastuzumab; Drug: Pertuzumab; Drug: taxane drug

INTERVENTIONS:
Drug: disitamab vedotin — disitamab vedotin 2mg/kg iv q2w
  Other Names: RC-48
  Arms: disitamab vedotin in combination with pyrotinib
Drug: Pyrotinib — pyrotinib 400mg po q28d
  Arms: disitamab vedotin in combination with pyrotinib
Drug: trastuzumab — trastuzumab 8mg/kg for the first cycle, 6mg/kg for subsequent treatments iv q21d
Drug: Pertuzumab — pertuzumab 840mg for the first cycle, 420mg for subsequent treatments iv q21d
  Arms: taxane drug in combination with trastuzumab and pertuzumab
Drug: taxane drug — Docetaxel/paclitaxel/albumin paclitaxel/liposomal paclitaxel, dosage and administration are determined according to the latest version of the NCCN and CSCO breast cancer guideline recommendations
  Arms: taxane drug in combination with trastuzumab and pertuzumab

SUMMARY:
The goal of this multicentre, randomized, double-blind controlled, phase III clinical trial is to compare the efficacy and safety of disitamab vedotin in combination with pyrotinib versus the standard first-line treatment of paclitaxel in combination with trastuzumab and pertuzumab (THP) for newly diagnosed recurrent/metastatic Human epidermal growth factor receptor 2 (HER2) positive advanced breast cancer, and to explore the impact of biomarkers on clinical efficacy and safety. The main questions it aims to answer are:

* Analyse the efficacy and safety of disitamab vedotin in combination with pyrotinib versus the standard first-line treatment of THP.
* Explore the impact of biomarkers on clinical efficacy and safety of the combination of disitamab vedotin in combination with pyrotinib treatment.

Participants in the experimental group will receive disitamab vedotin in combination with pyrotinib for 6-8 cycles (each cycle lasting 28 days), followed by maintenance treatment with trastuzumab in combination with pyrotinib. Participants in the control group will receive paclitaxel in combination with trastuzumab and pertuzumab for 6-8 cycles (each cycle lasting 21 days), followed by maintenance treatment with trastuzumab and pertuzumab.

Researchers will compare disitamab vedotin in combination with pyrotinib versus the standard first-line treatment of paclitaxel in combination with trastuzumab and pertuzumab to see if disitamab vedotin in combination with pyrotinib could be a new option for first-line treatment of HER2-positive metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Adult female patients (age 18-75 years) with metastatic breast cancer confirmed by pathology or imaging;
2. Pathologically confirmed HER2 positive (definition: Immunohistochemistry(IHC) 3+, or IHC 2+ and Fluorescent In Situ Hybridization(FISH) amplification);
3. No previous chemotherapy regimen for metastatic breast cancer;
4. At least one measurable lesion exists (Response Evaluation Criteria in Solid Tumors(RECIST) 1.1);
5. Eastern Cooperative Oncology Group(ECOG) performance status score ≤ 2 and expected survival of not less than 3 months;
6. Prior treatment-related toxicity at enrollment must have resolved to National Cancer Institute(NCI) Common Terminology Criteria for Adverse Events(CTCAE) (version 5.0) ≤ 1 degree (except for alopecia or other toxicity that, in the judgment of the investigator, is not considered a risk to the safety of the patient);
7. Patients with adequate organ function before enrollment:

   1. White Blood Cell (WBC) ≥ 3.0 x 10^9/L;
   2. Neutrophil granulocyte (ANC) ≥1.5 x 10^9/L;
   3. Platelet (PLT) ≥70×10^9/L;
8. Liver, kidney, and cardiac function tests are essentially normal (based on the normal values in the laboratory of each study center):

   1. Total bilirubin (TBIL) ≤ 3 x Upper Limit of Normal (ULN);
   2. Alanine aminotransferase (ALT/AST) ≤ 2.5 x ULN (≤ 5 x ULN in patients with liver metastases);
   3. serum creatinine ≤ 1.5 x ULN or creatinine clearance (Ccr) ≥ 60 ml/min;
9. . Normal cardiac function;

   1. Left ventricular ejection fraction (LVEF) ≥ 55%;
   2. QT-interval corrected with Fridericia (QTcF) ≤ 470ms;
10. Hormone receptor status is clear;
11. Female patients of childbearing potential who have a negative pregnancy test and agree to use an effective non-hormonal method of contraception during treatment and for at least 6 months after the last dose of the test drug;
12. Able to understand the study process, voluntarily participate in this study, and sign an informed consent form.

Exclusion Criteria:

1. Pathology suggestive of HER2 negativity (IHC 2+ and FISH-, or IHC 1+);
2. Patients with known hypersensitivity to the active ingredient or other components of the study drug;
3. Patients during pregnancy or lactation, patients with childbearing potential tested positive in a baseline pregnancy test, or patients unwilling to take effective contraceptive measures throughout the trial;
4. Patients not eligible for this study judged by the investigator, a pre-existing disease or condition that may interfere with participation in the study or any serious medical disorder that may interfere with the safety of the subject (e.g., uncontrolled heart disease, high blood pressure, active or uncontrolled infections, active hepatitis B virus infection).

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2023-09-06 (Actual); Primary Completion 2031-06-30 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Estimated 30 months
  From enrollment to progression or death (for any reason)

SECONDARY OUTCOMES:
Overall Survival (OS) | Estimated 8 years
  From enrollment to death (for any reason)
Disease control rate (DCR) | Estimated 30 months
  Ratio of complete response (CR) , partial response (PR) and stable disease (SD) in all subjects
Objective Response Rate (ORR) | Estimated 30 months
  Ratio of CR and PR in all subjects
Clinical Benefit rate (CBR) | Estimated 30 months
  Ratio of CR,PR and SD greater than or equal to 24 weeks in all subjects
Adverse Events (Based on CTCAE 5.0 standards) | From informed consent through 28 days following treatment completion
  Safety
Quality of Life (QoL) by Functional Assessment of Cancer Therapy for Breast Cancer (FACT-B) | Estimated 30 months
  QoL was assessed using FACT-B. FACT-B is a 37-item questionnaire with 5 subscales assessing physical, social, emotional, and functional well-being, with scores ranging from 0 to 4 for each question. Higher scores generally indicating a better quality of life.
Exploration of biomarkers | Estimated 30 months
  Next Generation Gene Sequencing (NGS) detection of tissue and blood specimens, including ERBB1/ERBB2/ERBB3/ERBB4/AKT/TP53/PIK3CA and so on. Objective to explore the correlation between biomarkers and the objective response rate (ORR), as well as progression-free survival (PFS).

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital,Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koleva-Kolarova RG, Oktora MP, Robijn AL, Greuter MJW, Reyners AKL, Buskens E, de Bock GH. Increased life expectancy as a result of non-hormonal targeted therapies for HER2 or hormone receptor positive metastatic breast cancer: A systematic review and meta-analysis. Cancer Treat Rev. 2017 Apr;55:16-25. doi: 10.1016/j.ctrv.2017.01.001. Epub 2017 Feb 20. PMID 28288388
- [Background] Mendes D, Alves C, Afonso N, Cardoso F, Passos-Coelho JL, Costa L, Andrade S, Batel-Marques F. The benefit of HER2-targeted therapies on overall survival of patients with metastatic HER2-positive breast cancer--a systematic review. Breast Cancer Res. 2015 Nov 17;17:140. doi: 10.1186/s13058-015-0648-2. PMID 26578067
- [Background] Wolff AC, Hammond MEH, Allison KH, Harvey BE, Mangu PB, Bartlett JMS, Bilous M, Ellis IO, Fitzgibbons P, Hanna W, Jenkins RB, Press MF, Spears PA, Vance GH, Viale G, McShane LM, Dowsett M. Human Epidermal Growth Factor Receptor 2 Testing in Breast Cancer: American Society of Clinical Oncology/College of American Pathologists Clinical Practice Guideline Focused Update. J Clin Oncol. 2018 Jul 10;36(20):2105-2122. doi: 10.1200/JCO.2018.77.8738. Epub 2018 May 30. PMID 29846122
- [Background] Swain SM, Miles D, Kim SB, Im YH, Im SA, Semiglazov V, Ciruelos E, Schneeweiss A, Loi S, Monturus E, Clark E, Knott A, Restuccia E, Benyunes MC, Cortes J; CLEOPATRA study group. Pertuzumab, trastuzumab, and docetaxel for HER2-positive metastatic breast cancer (CLEOPATRA): end-of-study results from a double-blind, randomised, placebo-controlled, phase 3 study. Lancet Oncol. 2020 Apr;21(4):519-530. doi: 10.1016/S1470-2045(19)30863-0. Epub 2020 Mar 12. PMID 32171426
- [Background] Glockner S, Buurman H, Kleeberger W, Lehmann U, Kreipe H. Marked intratumoral heterogeneity of c-myc and cyclinD1 but not of c-erbB2 amplification in breast cancer. Lab Invest. 2002 Oct;82(10):1419-26. doi: 10.1097/01.lab.0000032371.16521.40. PMID 12379776
- [Background] Shin SJ, Hyjek E, Early E, Knowles DM. Intratumoral heterogeneity of her-2/neu in invasive mammary carcinomas using fluorescence in-situ hybridization and tissue microarray. Int J Surg Pathol. 2006 Oct;14(4):279-84. doi: 10.1177/1066896906293055. PMID 17041191
- [Background] Brunelli M, Manfrin E, Martignoni G, Miller K, Remo A, Reghellin D, Bersani S, Gobbo S, Eccher A, Chilosi M, Bonetti F. Genotypic intratumoral heterogeneity in breast carcinoma with HER2/neu amplification: evaluation according to ASCO/CAP criteria. Am J Clin Pathol. 2009 May;131(5):678-82. doi: 10.1309/AJCP09VUTZWZXBMJ. PMID 19369627
- [Background] Cortes J, Kim SB, Chung WP, Im SA, Park YH, Hegg R, Kim MH, Tseng LM, Petry V, Chung CF, Iwata H, Hamilton E, Curigliano G, Xu B, Huang CS, Kim JH, Chiu JWY, Pedrini JL, Lee C, Liu Y, Cathcart J, Bako E, Verma S, Hurvitz SA; DESTINY-Breast03 Trial Investigators. Trastuzumab Deruxtecan versus Trastuzumab Emtansine for Breast Cancer. N Engl J Med. 2022 Mar 24;386(12):1143-1154. doi: 10.1056/NEJMoa2115022. PMID 35320644
- [Background] Modi S, Jacot W, Yamashita T, Sohn J, Vidal M, Tokunaga E, Tsurutani J, Ueno NT, Prat A, Chae YS, Lee KS, Niikura N, Park YH, Xu B, Wang X, Gil-Gil M, Li W, Pierga JY, Im SA, Moore HCF, Rugo HS, Yerushalmi R, Zagouri F, Gombos A, Kim SB, Liu Q, Luo T, Saura C, Schmid P, Sun T, Gambhire D, Yung L, Wang Y, Singh J, Vitazka P, Meinhardt G, Harbeck N, Cameron DA; DESTINY-Breast04 Trial Investigators. Trastuzumab Deruxtecan in Previously Treated HER2-Low Advanced Breast Cancer. N Engl J Med. 2022 Jul 7;387(1):9-20. doi: 10.1056/NEJMoa2203690. Epub 2022 Jun 5. PMID 35665782
- [Background] Yao X, Jiang J, Wang X, Huang C, Li D, Xie K, Xu Q, Li H, Li Z, Lou L, Fang J. A novel humanized anti-HER2 antibody conjugated with MMAE exerts potent anti-tumor activity. Breast Cancer Res Treat. 2015 Aug;153(1):123-33. doi: 10.1007/s10549-015-3503-3. Epub 2015 Aug 8. PMID 26253944
- [Background] Ocana A, Amir E, Pandiella A. HER2 heterogeneity and resistance to anti-HER2 antibody-drug conjugates. Breast Cancer Res. 2020 Jan 31;22(1):15. doi: 10.1186/s13058-020-1252-7. PMID 32005279
- [Background] Rios-Doria J, Harper J, Rothstein R, Wetzel L, Chesebrough J, Marrero A, Chen C, Strout P, Mulgrew K, McGlinchey K, Fleming R, Bezabeh B, Meekin J, Stewart D, Kennedy M, Martin P, Buchanan A, Dimasi N, Michelotti E, Hollingsworth R. Antibody-Drug Conjugates Bearing Pyrrolobenzodiazepine or Tubulysin Payloads Are Immunomodulatory and Synergize with Multiple Immunotherapies. Cancer Res. 2017 May 15;77(10):2686-2698. doi: 10.1158/0008-5472.CAN-16-2854. Epub 2017 Mar 10. PMID 28283653
- [Background] Li BT, Michelini F, Misale S, Cocco E, Baldino L, Cai Y, Shifman S, Tu HY, Myers ML, Xu C, Mattar M, Khodos I, Little M, Qeriqi B, Weitsman G, Wilhem CJ, Lalani AS, Diala I, Freedman RA, Lin NU, Solit DB, Berger MF, Barber PR, Ng T, Offin M, Isbell JM, Jones DR, Yu HA, Thyparambil S, Liao WL, Bhalkikar A, Cecchi F, Hyman DM, Lewis JS, Buonocore DJ, Ho AL, Makker V, Reis-Filho JS, Razavi P, Arcila ME, Kris MG, Poirier JT, Shen R, Tsurutani J, Ulaner GA, de Stanchina E, Rosen N, Rudin CM, Scaltriti M. HER2-Mediated Internalization of Cytotoxic Agents in ERBB2 Amplified or Mutant Lung Cancers. Cancer Discov. 2020 May;10(5):674-687. doi: 10.1158/2159-8290.CD-20-0215. Epub 2020 Mar 25. PMID 32213539